CLINICAL TRIAL: NCT06999954
Title: The Shwachman-Diamond Syndrome Global Patient Survey and Partnering Platform Program (SDS-GPS Program)
Brief Title: Shwachman-Diamond Syndrome Global Patient Survey and Partnering Platform
Acronym: SDS-GPS
Status: Recruiting | Type: Observational
Sponsor: Shwachman-Diamond Syndrome Alliance Inc (Other)
Responsible Party: Sponsor
Other Study IDs: NB300118
Record Dates: First submitted 2024-07-20; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Shwachman-Diamond Syndrome; SDS; IBMF; Congenital Neutropenia; Heme Malignancy; Shwachman Syndrome; Inherited Bone Marrow Failure; Exocrine Pancreatic Insufficiency; WHIM; ELANE; SBDS Gene Mutation; EFL1 Gene Mutation; DNAJC21 Gene Mutation; SRP54 Gene Mutation; Inherited Cancer Syndrome; Inherited Cancer-Predisposing Syndrome; Neutropenia, Severe Chronic; Neutropenia Other; Neutropenia Chronic Benign; Ribosome Alteration; Ribosomopathy; Immune Deficiency; Inherited BMF Syndrome; Inherited Immunodeficiency Diseases; Cognitive Delay, Mild; Myelodysplastic Syndromes; Pancytopenia
Keywords: Shwachman-Diamond Syndrome; Shwachman Diamond Syndrome; Shwachman Syndrome; SDS; IBMF; Inherited Bone Marrow Failure; Congenital Neutropenia; Immune Deficiency; SDS-like syndrome; genetic cancer predisposition; WHIM; ELANE; SBDS; EFL1; SRP54; DNAJC21; severe chronic neutropenia; exocrine pancreatic insufficiency; ribosomopathy
MeSH Terms: conditions — Shwachman-Diamond Syndrome; Neutropenia, Severe Congenital, Autosomal Recessive 3; Exocrine Pancreatic Insufficiency; Neoplastic Syndromes, Hereditary; Neutropenia, severe chronic; Immunologic Deficiency Syndromes; Congenital Bone Marrow Failure Syndromes; Primary Immunodeficiency Diseases; Lymphoma, Follicular; Myelodysplastic Syndromes; Pancytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 120 Years
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The Shwachman-Diamond Syndrome Global Patient Survey and Collaboration Program (SDS-GPS) is an opportunity for patients and their families - from anywhere in the world - to share their experience living with SDS via a safe, secure, and convenient online platform, to

* expand the understanding of SDS
* improve the lives of people with SDS, and
* accelerate the development of new therapies and cures for SDS.

By joining, participants will receive early access to relevant information about new clinical trials and other research opportunities (such as clinical registries) based on their profile, accelerating research and increasing clinical trial impact and recruitment success.

The platform, consent forms, and surveys are available in five languages: English, Spanish, French, German, and Italian. More languages to come.

DETAILED DESCRIPTION:
What is SDS-GPS?

The Shwachman-Diamond Syndrome Global Patient Survey and Collaboration Program (SDS-GPS) is an opportunity for patients and their families - from anywhere in the world - to share their experience living with SDS via a safe, secure, and convenient online platform, with the goal of

* expanding the understanding of SDS and related conditions
* improving the lives of people with SDS and related conditions, and
* accelerating the development of new therapies and cures for SDS.

SDS-GPS was created for the patients, by the patients, with thoughtful input from patients, families, advocates, caregivers, researchers, clinicians, and regulators.

Participants will be part of a global community that cares, turns hope into action, and drives research. Participants' experience - whether it falls in the mild or severe end of the spectrum - matters. Their voice counts.

How can patients' stories help drive therapies and cures?

Participants' stories help paint a more complete picture of what SDS is and how it impacts the people living with it. Their participation helps build a strong, engaged community, which is critical to drive progress. Without patients and their families, research cannot advance.

The investigators (the SDS-GPS team at the SDS Alliance) use participants' de-identified aggregate survey responses and other data they share to develop a deeper understanding of the unmet needs of the community.

The investigators use the insights to

* Prioritize research, educational resources, and community programming
* Promote data and knowledge sharing via collaborations, publications, conference presentations, and other communication channels
* Provide participants with information about relevant research opportunities (such as the SDS Registry and other natural history studies), clinical trials, educational resources, and community support connections.

What aspects of their story can participants share through SDS-GPS?

Surveys on the SDS-GPS Program Platform are designed to be quick and easy, without the need to have to look up any details from medical records. They can save their progress and come back anytime.

Survey topics include:

* Socio-demographics
* Medical history and diagnostics
* Treatment and disease progression
* Management of and access to care
* Quality of life

How does SDS-GPS work?

* Sign up for a free SDS-GPS account and enter a little bit about the participant. Enrolling and participating takes little time, and they can come back later to update any information.
* Answer surveys from the comfort of their home at any time that works for them.
* Privacy and security are protected to the highest standard.
* Move research forward without any clinic visits or virtual appointments. With participants' consent, the investigators publish and share de-identified data (your survey responses) with approved researchers to support research to benefit the SDS community. The information participants provide through easy surveys is structured and coded behind the scenes, to be usable for high-quality, impactful research.
* Keep track of the participants' medical appointments, medications, and symptoms via their SDS-GPS account, and have all the information at their fingertips whenever and wherever they need it.
* Share any information participants like with their care team. Participants retain full control over access.

The platform, consent forms, and surveys are available in five languages: English, Spanish, French, German, and Italian. More languages to come.

ELIGIBILITY:
Inclusion Criteria:

The Program invites patients of all ages who have a confirmed diagnosis of the below, using established diagnostic guidelines, plus their parents/caregivers.

* Patients with a confirmed Shwachman-Diamond Syndrome (SDS) diagnosis, including a genetic or clinical diagnosis. The initial focus will be on patients with a genetic diagnosis of SDS based on biallelic mutations in SBDS or EFL1.
* Patients with a confirmed diagnosis of an SDS-like syndrome (e.g. due to mutations in DNAJC21, SRP54, or other genes that may be associated with an SDS-like syndrome in the future).
* Patients with other heritable hematological malignancy disorders (such as RUNX1-FPD, Fanconi Anemia) and/or congenital neutropenias (such as ELANE neutropenia) are also eligible for inclusion.
* Caregivers, parents, and close relatives of all patients above, including of patients alive or deceased.

Exclusion Criteria:

● People who do not meet the above criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients and their caregivers may enroll from anywhere in the world using our online platform. Individuals for whom English is not their primary language may be enrolled with a translated informed consent form (and translated surveys if available). Currently available languages include English, Spanish, French, Italian, and German.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2088-12 (Estimated); Study Completion 2088-12 (Estimated)

PRIMARY OUTCOMES:
Patient (or caregiver) reported symptoms over time | At baseline and every 12 months, prospectively.
  Patients report symptoms via surveys, grouped by organ system.
Genetics report uploaded by patient (or caregiver) | Through study completion when the genetics report is available.
  Clinical genetics reports are uploaded by the patient (or caregiver) and curated by study staff to confirm a genetic diagnosis, understand variants, and assess the use of appropriate genetic testing methodologies.
Quality of life measures via PROMIS surveys | Through study completion, an average of 2-4 times per year.
  PROMIS surveys in various domains, such as fatigue, pain, anxiety, and depression, are administered as surveys and scored with the standard PROMIS scoring methods.
  Specific PROMIS measures to include:
  v1.0 Anxiety 8a short form v1.0 Depression 8a short form v1.0 Pain Interference 6a short form v2.0 Cognitive Function 8a short form v1.0 Self-Efficacy for Managing Chronic Conditions: Manage Daily Activities 8a short form v1.0 - Self-Efficacy for Managing Symptoms 8a v2.0 Satisfaction Social Roles and Activities 8a short form v2.0 Ability to Part Social Roles and Activities 8a short form v2.0 Social Isolation 8a short form v1.0 Fatigue 13a short form (FACIT-Fatigue)
  v3.0 PP: Depressive Symptoms 6a short form v3.0 PP: Fatigue 10a short form v3.0 PP: Mobility 7a short form v3.0 PP: Pain Interference 8a short form v1.0 PP: Cognitive Function 7a short form
Patient reported burden of disease and treatment outcomes | At baseline and every 12 months, prospectively.
  Patients fill out surveys to report on disease burden (such as number and duration of hospitalizations), treatment burden (such as surveillance), and treatment outcomes (such as HSC transplant outcomes)

CONTACTS AND LOCATIONS:
Locations (1):
- Shwachman-Diamond Syndrome Alliance Inc., Woburn, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study is focused on patient reported data and findings will be published in the aggregate to safeguard patient personal health information.

REFERENCES:
- See also: General information page for participants, including frequently asked questions and answers. — https://www.sdsalliance.org/sds-gps
- Available data/document: Informed Consent Form — https://www.sdsalliance.org/sds-gps — Available from the SDS-GPS program team at gps@sdsalliance.org